CLINICAL TRIAL: NCT00564109
Title: Are the Pancreatic Serum Proteins Pancreatic Stone Protein (PSP) and Pancreatitis-Associated Protein (PAP) Predictive for the Development of Sepsis? Retrospective Study in Trauma Patients With Soft Tissue Defects.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Marius Keel, University Hospital Zurich
Other Study IDs: StV 10-2003
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2007-11

CONDITIONS: Trauma Patients With Soft Tissue Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: retrospective Observation — retrospective Observation

SUMMARY:
Retrospective analysis of PSP- and PAP-serum levels in trauma patients with soft tissue defects and possible correlation with the incidence and onset of infection and sepsis.

ELIGIBILITY:
Inclusion criteria:

* Trauma patients submitted to the university hospital Zurich, aged 18-65 with soft tissue defects

Exclusion criteria:

* Patients with known immunocompromising illnesses, drug abuse or infectious diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2005-08; Study Completion 2008-01

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland